CLINICAL TRIAL: NCT00677911
Title: Immunologic Response to Negative Cognition in Persons With Chronic Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: American Pain Society (Other)
Responsible Party: Principal Investigator, Beth Darnall, PhD, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Purpose: Other
Other Study IDs: OCTRI975
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Interleukin-6; pain catastrophizing; cytokines; cortisol
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: In-vivo pain catastrophizing induction — All participants underwent a 10-minute in-vivo pain castastrophizing induction.

SUMMARY:
Principal Investigator/Program Director (Last, First, Middle): Darnall, Beth APS Future Leaders in Pain Small Research Grants Application Page 5 Continuation Format Page

Summary: Chronic pain is stressful, both physically and psychologically. Stressful experiences induce autonomic nervous system arousal, which reliably leads to inflammation and immune suppression. Inflammation then exacerbates existing pain and may be a key factor in both the genesis and maintenance of pain. Stress-induced immune effects are detected two hours (2 hrs) post-stressor, suggesting only a few stressful experiences per day may be sufficient to sustain elevated pain levels1. Cognition has emerged as a potential mediating factor in the relationship between pain and stress. Mentally recreating an emotionally stressful event induces de novo physiological stress1. In other words, thinking about an emotionally charged event down-regulates autonomic stress responses and subsequent immune effects. Therefore, exploring cognition as a mediating factor between stress, pain, and inflammation will inform our understanding of pain pathways, as well as improve treatment for pain.

Study Rationale: The acute stress response induces immunosuppression; however, this relationship has been studied in arbitrary models only (shock avoidance, job interview). This study employs the novel approach of examining stress and immune responses to a personally relevant stressor (pain); prior studies used arbitrary models only (shock avoidance, job interview). Pain offers a highly salient and personal context well-suited for investigation of negative cognitive perseveration. Pain is acutely sensitive to exacerbation via inflammation, and thus the relevance of examining immune effects of rumination on future negative expectations ("expecting the worst") is underscored.

Goal: To test the biological consequences of negative expectations, achieved via an active 10-minute negative cognitive perseveration on a personally relevant stressor: future worsening of one's chronic pain condition. Biological stress response will be measured via heart rate (HR), blood pressure (BP) and serum cortisol. Impact of negative cognition on inflammation will be measured using interleukin-1 (IL-1), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) as biomarkers of immune function, controlling for depression and pain catastrophizing. This study aims to inform the understanding of pain mechanisms.

Aim 1: Determine the magnitude of an autonomic stress response to an induction of negative cognition.

Aim 2: Determine immune effects of the experiment-induced stress response.

Aim 3: Establish whether a pre-existing tendency to catastrophize mediates the relationship between experiment-induced negative perseveration and immune effects.

Aim 4: Establish whether stress-related increases in IL-6 remain elevated post 2 hrs.

DETAILED DESCRIPTION:
Methods: This prospective study examines the magnitude of biological stress and subsequent immunologic changes in response to negative cognitive perseveration. Five physiological measurement time points occur over the course of the 3 hour experiment.

Demographics and health characteristics of interest: gender, marital status, smoking status, education level, race, height, weight, body mass index, medical comorbidity, psychological comorbidity, medications (for inflammation, pain, or psychiatric conditions).

Inclusionary Criteria

* >18 years of age; <65 years of age
* Non-inflammatory musculoskeletal patients presenting for evaluation at Oregon Health & Science University (OHSU) Comprehensive Pain Center (CPC)

Exclusionary Criteria

* Active or recent virus/infection
* Thought disorder, Suicidality,
* Substance Abuse
* Active corticosteroid regimen
* Pregnancy
* Limited venous access
* Former intravenous drug user

Enrollment: All persons presenting for evaluation at the CPC who meet study criteria will be offered the option to participate in the study. Approximately 60 new pain patients are evaluated by psychology monthly and we expect to obtain our goal of 40 participants within 6 months. Informed consent will be obtained in compliance with OHSU Institutional Review Board protocol. Subjects will receive $100 gift certificate compensation, even if they fail to complete the study. We anticipate a low completion failure rate as the study is completed in one 3-hour time block. Study times will be standardized to account for circadian effects. Participants will be told to arrive having eaten a light breakfast with minimal caffeine consumption (e.g., less than 2 cups of coffee). They will be given a subject number and their psychiatric diagnoses will be blinded to prevent bias. The study involves gathering 5 serum samples and thus participants will be catheterized by nursing staff to minimize physiological stress.

Principal Investigator/Program Director (Last, First, Middle): Darnall, Beth APS Future Leaders in Pain Small Research Grants Application Page 7 Continuation Format Page

Study site: The study will be conducted at the NIH-funded General Clinical Research Center (GCRC). The GCRC provides state of the art resources including research space, specialized research nurses to perform blood draws and gather biodata, biostatisticians, and sophisticated laboratories to perform serum biomarker analysis. OHSU's GCRC is Oregon's premier multidisciplinary patient-oriented research facility and is housed in the same building as the CPC, thus minimizing travel burden on participants.

Active Stress Induction: Negative Cognitive Perseveration On their experiment day, participants will interface with a licensed clinical psychologist who did not perform their clinical interview and who is blinded to their diagnoses. The psychologist will instruct the participant talk for 10 minutes about the worst aspects of their pain, to discuss their loss of control over their situation, the negative impact pain has had on their life and others. They will be guided to imagine that their situation will progressively worsen, and to focus on how badly they will feel as a result. Two measures of induction efficacy will be given: subjective verbal rating (0-10) and objective rating by attending psychologist (0-10). The intervention ends at 10 minutes and the remainder of the study involves biodata measurement.

Study ends at 2.5 hrs post induction following the final blood draw. The psychologist will debrief subjects and will assess their affective state. Their subjective units of distress will be checked. Persons who are in a continued negative cognitive state will receive 30 minutes of Cognitive Behavioral Therapy (CBT) by the on-site psychologist. Care will be taken not to allow participants to leave the study site in distress. Participants will receive follow up psychology care at the CPC as indicated in their treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* chronic musculoskeletal pain
* being treated for chronic pain at OHSU

Exclusion Criteria:

* suicidality or thought disorder
* pregnant
* poor venous access
* current corticosterioid regimen
* recent or active virus or infection
* substance abuse
* former IV drug user

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 | cross-sectional

CONTACTS AND LOCATIONS:
Locations (1):
- OCTRI; OHSU Mail Code: CHH 13th floor 3303 Bond St., Portland, Oregon, United States